CLINICAL TRIAL: NCT03242993
Title: Biodistribution, Tumor Detection, and Radiation Dosimentry of [18F]-AZAFOL as POSITRON EMISSION TOMOGRAPHY (PET) Tracer in Folate Receptor Positive Cancer Imaging
Brief Title: [18F]-AZAFOL AS POSITRON EMISSION TOMOGRAPHY (PET) TRACER in FR Positive Cancer Imaging
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Lausanne Hospitals (Other)
Collaborators: University Hospital, Zürich (Other); Cantonal Hospital of St. Gallen (Other)
Responsible Party: Principal Investigator, Niklaus Schaefer, clinical professor, University of Lausanne Hospitals
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PET - FOL - I
Record Dates: First submitted 2017-07-20; First posted 2017-08-08 (Actual); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Metastatic Cancer Lung; Metastatic Ovarian Cancer
MeSH Terms: conditions — Lung Neoplasms; Ovarian Neoplasms | interventions — Folic Acid

STUDY DESIGN:
Intervention Model Description: This is a single arm study. No placebo or other comparator will be used. [18F]-AzaFol is used as a PET tracer, all patients successfully enrolled will be assigned to the treatment group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment group (Experimental): all patients successfully enrolled will be assigned to the treatment group:
  1 mg folic acid (corresponding to 0.2 mL Folarell®) will be injected 5 min prior to [18F]-AzaFol
  Interventions: Drug: [18F]-AzaFol; Drug: folarell

INTERVENTIONS:
Drug: [18F]-AzaFol — [18F]-AzaFol is a radiotracer produced at ETH Hönggerberg in a radiopharmaceutical GMP facility. The drug product is provided as sterile solution for intravenous injection in a glass vial containing 6 mL of formulated product, the maximal applicable dose being 600 MBq.
Drug: folarell — For the purpose of this study only 1 mg folic acid (corresponding to 0.2 mL Folarell®) will be injected 5 min prior to [18F]-AzaFol. Due to this low dose of a single injection of folic acid it is unlikely that adverse events would occur.
  Folarell® is a folic acid preparation for intravenous or intramuscular injection
  Other Names: folic acid

SUMMARY:
This is a clinical trial category C as this is a first in man trial with an unapproved investigational product. Nevertheless the risk is considered low due to the low dose ≤ 10μg. No toxicity effects were observed preclinically at a dose >1000 -fold the intended dose. Open-labeled, non-blinded, non-placebo controlled, multicenter study.

Primary objective:

Assessment of biodistribution and FR-specific tumor detection of [18F]- AzaFol as a PET imaging agent in patients with FR-positive and FR-negative metastatic cancer of the ovaries or lungs.

Secondary objective:

Calculation of the effective dose to the patient according to the tissue distribution data of [18F]-AzaFol (Dosimetry)

DETAILED DESCRIPTION:
Human research study using a radiopharmaceutical product to reveal folate receptor (FR) expression in tumors in patients.

It is known that the FR is overexpressed on a variety of tumor types. FR-positive tumors can be treated with investigational drugs specifically targeting the FR.

Although the FR-expression status may be determined by immunohistochemical staining of tumor biopsies there is a need for a non-invasive method to determine the presence of the FR on primary tumors and metastases in humans. For this purpose a radiopharmaceutical product will be used as a radiotracer. Positron Emission Tomography (PET) is an imaging method which allows assessing the distribution of radiotracers (called PET tracer). With this imaging method it is possible to obtain (semi)quantitative measures of FR-expression on tumors of at least 4-10 mm diameter in patients.

Such a folate-based radiotracer would be a very helpful tool to non-invasively discriminate FR-positive (often found in ovarian and NSC-lung cancer) from FR-negative tumors in patients with cancer disease as this would allow selecting FR-positive patients amenable to FR-targeted therapies, e.g. folate-targeted antimitotic substances such as EC145 VintafolideTM (Endocyte Inc.) or anti-FR-antibodies such as FarletuzumabTM (Morphotek Inc).

Moreover, [18F]-AzaFol PET could be used for tumor staging and monitoring therapy as well as for follow-up investigations of patients with FR-positive tumors.

Currently there is a radiopharmaceutical product for research purposes available (99mTc-EC20, EtarfolatideTM, Endocyte Inc.) which can be used for Single Photon Emission Computed Tomography (SPECT) imaging. SPECT, however, has multiple limitations compared to PET, such as inferior spatial resolution, soft tissue attenuation, lack of dynamic acquisition etc. Therefore, a PET-compound for FR imaging has been shown to image FR-positive tumors in experimental animals .

Calculations regarding the incidence and mortality of six frequent cancer types in Switzerland indicate that in over 53% of the new cases the FR is expressed (OncoSuisse, Cancer Statistics 2012).

Investigators demonstrate impressively why FR-targeting emerged as an attractive strategy for tumor diagnosis and for the development of new targeted therapy strategies .

The vitamin folic acid (pteroylglutamic acid) emerged as an almost ideal FR-targeting agent because of the high affine binding to the FR (KD < 1 nM).

Due to the small size and vitamin character of folic acid, it is non-immunogenic and non-toxic.

In spite of a large number of folate-based nuclear imaging agents which have been developed in the last two decades only one SPECT radiotracer (99mTc-EC20, EtarfolatideTM) is currently being used in clinical trials in the U.S. for SPECT imaging. For over a decade investigators have been focusing research activities on the development of a 18F-based folate radiotracer for PET imaging (13-16). Recently, a novel folate radiotracer has been developed, 3'-aza-3-[18F]fluorofolic acid (herein referred to as [18F]-AzaFol), for PET imaging purposes.

Compared to SPECT, PET is the more sensitive nuclear imaging method which provides images of an improved resolution and the possibility for accurate quantification of accumulated radioactivity in tumor lesions.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cancer of the ovaries (adenocarcinoma) or non-small cell lung cancer (adenocarcinoma, squameous cell cancer or other histology) having active tumor with an indication for a systemic treatment in first or further line.
* Last systemic treatment should not applied within 3 weeks before performing study exam
* Male and female patients 18 years and older,
* Voluntarily signed Informed Consent after being informed

Inclusion criteria for [18F]-AzaFol PET (enrollment into study):

* FR-positive histology in routinely acquired biopsy samples (30 Patients)
* FR-negative histology in routinely acquired biopsy samples (6 Patients)

Exclusion Criteria:

* contraindications to the class of drugs under study, e.g. known hypersensitivity or allergy to class of drugs or the investigational product,
* women who are pregnant or breast feeding,
* women with the intention to become pregnant during the course of the study,
* other clinically significant concomitant disease states (e.g., renal failure, hepatic dysfunction, cardiovascular disease),
* Renal clearance < 60 mL/min; liver transaminases ≥ 3-fold increased; bilirubin > 1.5-fold increased; Hb < 8 g/dl; Tc < 100'000, ANC < 1'500/ul
* ECOG 3-4
* known or suspected non-compliance, drug or alcohol abuse,
* inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the subject,
* Participation in another study with an investigational drug during the present study and 7 days thereafter.
* Enrolment of the investigator, his family members, employees and other dependent persons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
SUV values and volume of tracer uptake of all suspected positive lesions | day 0
  SUVmax g/ml SUVmean42% g/ml
  lesion seen on SOC : mm
Potential change of overall staging | day 0
  TNM staging
Lesion detection rate in comparison to SOC (CT and/or MR and/or FDG performed within 4 weeks of PET imaging). | day 0
  % (percentage)
Estimation of gained information using this tracer | day 0
  uptake yes / no
quantitative estimations | day 0
  SUV values for ROC analysis g/ml
General estimation of gained confidence in changing/adapting therapy based on this image | day 0
  continuous % variable of confidence
Available biopsy results can be used as further variables to better assess the performance of [18F]-AzaFol | day 0
  + / - ( positive or negative)

SECONDARY OUTCOMES:
Calculation of the effective dose to the patient according to the tissue distribution data of [18F]-AzaFol (Dosimetry) | day 0
  The secondary outcome is the calculated tissue distribution data of [18F]-AzaFol obtained in humans. The effective dose for all organs will be calculated using the OLINDA software (version 1.0). The data will be compared to the estimated data from our preclinical data set. This will provide the radiation dosimetry values as well as quantitative biodistribution over all relevant organs.

CONTACTS AND LOCATIONS:
Overall Officials: John Prior, Prof, Principal Investigator — Lausanne University Hospitals
Locations (1):
- Lausanne University Hospitals, Lausanne, Canton of Vaud, Switzerland

REFERENCES:
- [Derived] Gnesin S, Muller J, Burger IA, Meisel A, Siano M, Fruh M, Choschzick M, Muller C, Schibli R, Ametamey SM, Kaufmann PA, Treyer V, Prior JO, Schaefer N. Radiation dosimetry of 18F-AzaFol: A first in-human use of a folate receptor PET tracer. EJNMMI Res. 2020 Apr 8;10(1):32. doi: 10.1186/s13550-020-00624-2. PMID 32270313